CLINICAL TRIAL: NCT02450591
Title: Pilot Study of Local Therapies for Oligometastatic Non-Small Cell Lung Cancer Harboring Sensitizing EGFR Mutations
Brief Title: Local Therapies for Oligometastatic Non-Small Cell Lung Cancer Harboring Sensitizing EGFR Mutations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-067
Record Dates: First submitted 2015-05-14; First posted 2015-05-21 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2017-12

CONDITIONS: Oligometastatic Lung Adenocarcinoma
Keywords: Sensitizing EGFR Mutations; Erlotinib; Surgery; Radiation Therapy; 15-067
MeSH Terms: interventions — Erlotinib Hydrochloride

ARMS (1):
- Oligometastatic Non-Small Cell Lung Cancer (Experimental): Patients will be placed on EGFR-TKI for their metastatic EGFR-mutant stage IV oligometastatic disease. All patients will undergo induction TKI for 12 weeks. At the conclusion of 12 weeks on erlotinib, patients without disease progression [partial response (PR) or stable disease (SD)] will undergo definitive local treatment to all remaining sites of disease. After local therapy, erlotinib will be resumed until progression of disease (POD) by RECIST criteria. All assessments completed during the 12 week TKI induction phase are to be performed per protocol with a ± 7 day window.
  Interventions: Drug: Erlotinib; Other: Local Therapies

INTERVENTIONS:
Drug: Erlotinib
Other: Local Therapies — Definitive local therapies include surgical resection, stereotactic radiosurgery, ablation and conventional radiation therapy

SUMMARY:
This study will test if local therapies in addition to erlotinib can improve responses and delay the time until new treatment is required. This study will also collect blood samples for research blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed metastatic lung adenocarcinoma (recurrent or de novo) harboring sensitizing EGFR mutations (L858R, exon 19 deletion, G719A, L861Q, S768I, exon 19 insertions) with oligometastatic disease (≤5 discrete lesions of disease irrespective of location, inclusive of the primary lesion):
* all sites of disease must be amenable to definitive treatment with a local therapy (surgical resection, stereotactic radiosurgery, ablation and conventional radiation therapy) as determined by surgery, interventional radiology and radiation oncology
* all intrathoracic lymph nodes (including hilar, mediastinal, and supraclavicular nodal disease) are considered 1 discrete lesion.
* Each brain metastasis is included as a distinct lesion.
* Patients already started on erlotinib are eligible as long as their sites of disease are determined to be eligible for definitive local therapy by consensus of the principal investigators within 12 weeks of the patient first taking erlotinib.
* Lung adenocarcinoma histology confirmed at MSKCC.
* Available archived tissue to perform molecular analysis
* Patients without available archived tissue can have repeat biopsies to determine EGFR status as per standard clinical care guidelines
* Age 18 years or older
* Karnofsky Performance Status ≥ 70%
* Adequate bone marrow, liver and renal function, as specified below:
* Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
* Hemoglobin ≥ 8 g/dL
* Platelets ≥ 100 x 109/L
* Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) (except for patients with documented Gilbert's Syndrome)
* AST and ALT ≤ 2.5 x ULN or ≤ 5 x ULN if liver metastases are present
* Serum creatinine ≤ 1.5 x upper limit of normal or creatinine clearance ≥ 60ml/min for patients with creatinine levels above institutional normal.
* For women of child-bearing potential, negative pregnancy test within 14 days prior to starting treatment
* Men and women of childbearing age must be willing to use effective contraception while on treatment and for at least 3 months thereafter

Exclusion Criteria:

* Treatment with erlotinib prior to developing metastatic disease
* Patients with activating but not sensitizing mutations (exon 20 insertions, EGFR T790M)
* Malignant pleural effusion or pleural disease
* Leptomeningeal disease
* Any site of disease that is not amenable to definitively local therapy including surgery or radiation therapy
* Women who are breastfeeding or pregnant
* Concurrent malignancies other than non-melanoma skin cancer that require active ongoing treatment.
* Any medical co-morbidities that would preclude surgery or radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oligometastatic Non-Small Cell Lung Cancer
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oligometastatic Non-Small Cell Lung Cancer
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 61 [55 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by at Least Five Patients Will Need to Complete Local Therapy.
Description: At least five patients will need to complete local therapy within 2 years of the study being open to accrual for the primary endpoint to be met.
Time Frame: 2 years
Population: Primary outcome accrual goal was not achieved. Data were not collected.
Arm/Group | Oligometastatic Non-Small Cell Lung Cancer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days (+/- 7 days) after treatment completion
Arm/Group | Oligometastatic Non-Small Cell Lung Cancer
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oligometastatic Non-Small Cell Lung Cancer (N=4)
Seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oligometastatic Non-Small Cell Lung Cancer (N=4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Blood bilirubin increased (Investigations) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Keratitis (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT02450591/Prot_SAP_000.pdf